CLINICAL TRIAL: NCT05691153
Title: A Single-center, Dose Selection Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Allogeneic CAR-T Targeting CD19 in Patients With Auto-CAR T Relapsed B-cell Non-Hodgkin's Lymphoma
Brief Title: ThisCART19A for B-NHL Relapsed After Auto-CAR T
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Fundamenta Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZ5602
Record Dates: First submitted 2022-12-27; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: CAR; B Cell Lymphoma; Relapsed Non-Hodgkin Lymphoma
Keywords: Universal CAR-T
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Level 1 (Experimental): ThisCART19A，2×10^6 cells/kg（Single dose of Allogeneic Anti-CD19 CAR T cells will be infused）
  Interventions: Drug: ThisCART19A with Dose Level 1
- Dose Level 2 (Experimental): ThisCART19A，3×10^6 cells/kg（Single dose of Allogeneic Anti-CD19 CAR T cells will be infused）
  Interventions: Drug: ThisCART19A with Dose Level 2

INTERVENTIONS:
Drug: ThisCART19A with Dose Level 1 — ThisCART19A，2×10^6 cells/kg（Single dose of Allogeneic Anti-CD19 CAR T cells will be infused）, after the lymphodepletion conditioning of fludarabine, CTX and VP-16
  Other Names: ThisCART19A with 2×10^6 cells/kg
  Arms: Dose Level 1
Drug: ThisCART19A with Dose Level 2 — ThisCART19A，3×10^6 cells/kg（Single dose of Allogeneic Anti-CD19 CAR T cells will be infused）, after the lymphodepletion conditioning of fludarabine, CTX and VP-16
  Other Names: ThisCART19A with 3×10^6 cells/kg
  Arms: Dose Level 2

SUMMARY:
This is a phase 1, single-center, dose selection study to evaluate the efficacy, safety, and pharmacokinetics of ThisCART19A (allogeneic CAR-T targeting CD19) in patients with Auto-CAR T relapsed B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
This is a phase 1, single-center, dose selection study to evaluate the efficacy, safety, and pharmacokinetics of ThisCART19A in patients with Auto-CAR T relapsed B-cell non-Hodgkin's lymphoma. The study will identify a treatment regimen most likely to result in clinical efficacy while maintaining a favorable safety profile. Before initiating ThisCART19A infusion, subjects will be administered lymphodepletion chemotherapy composed of fludarabine、cyclophosphamide and VP-16. At Day 0 of the Treatment Period, subjects will receive an intravenous (IV) infusion of ThisCART19A. All subjects are monitored during the treatment period through Day 28. All subjects who receive a dose of ThisCART19A will be followed up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a documented IRB-approved ICF prior to any screening procedure;
2. Gender not restricted, 18 years ≤ age ≤ 75 years;
3. Subjects with Auto-CAR T relapsed B-cell non-Hodgkin's lymphoma;
4. Life expectancy ≥ 12 weeks at the time of enrollment;
5. Eastern Cooperative Oncology Group performance status score of 0 or 1;
6. At least one measurable lesion to be assessed, with any nodal lesion > 15mm in LDi (longest diameter) and any extranodal lesion > 10mm in LDi;
7. Subject has adequate bone marrow, renal, hepatic, pulmonary, and cardiac function defined as:

   1. Adequate marrow function for lymphodepletion chemotherapy: 14 days before enrollment, absolute neutrophil count (ANC) ≥ 1×10^9/L, platelet count ≥ 30×10^9/L, hemoglobin ≥ 80 g/L without blood transfusion;
   2. Creatinine clearance ≥ 30 ml/min according to the Cockcroft-Gault formula, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × the upper limit of normal (ULN), total bilirubin ≤ 2×ULN (Subjects with Gilbert syndrome or liver involvement may be enrolled if their total bilirubin is ≤ 3×ULN);
   3. Pulmonary function: Baseline oxygen saturation (SaO2) ≥ 92% on room air;
   4. Cardiac function：left ventricular ejection fraction (LVEF) ≥ 40% assessed by echocardiography.
8. CD19-positive lymphoma confirmed on a biopsy during screening.

Exclusion Criteria:

1. Allergic to preconditioning measures in the trial.
2. Other malignancies apart from B-cell malignancies within 5 years prior to screening. (Subjects with cured skin squamous carcinoma, basal carcinoma, non-primary invasive bladder cancer, localized low-risk prostate cancer, in situ cervical/breast cancer can be recruited.)
3. Severe active infection (Simple urinary tract infection (UTI) and uncomplicated bacterial pharyngitis are permitted).
4. Pulmonary embolism (PE) within 3 months prior to enrollment.
5. Intolerant severe cardiovascular and cerebrovascular diseases and hereditary diseases assessed by the investigator prior to enrollment.
6. Gastrointestinal involvement at risk of active bleeding.
7. Massive pericardial effusion, symptomatic thoracic or abdominal effusion.
8. Presence of CNS involvement (both primary and secondary) at screening confirmed by imaging or CSF testing.
9. Active hepatitis B virus (serum HBV-DNA ≥ 2000 IU/mL), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or active syphilis infection prior to enrollment. (Patients with HBV-DNA < 2000 IU/mL can be enrolled, but should be administered antiviral drugs such as entecavir and tenofovir with relative clinical indicators monitored simultaneously during the treatment.)
10. Less than 100 days after allogeneic hematopoietic stem cell transplantation.
11. Vaccinated with influenza vaccine within 2 weeks prior to lymphodepletion chemotherapy. (Patients vaccinated with SARS-COV19 vaccine or inactivated; live/non-live adjuvant vaccines can be enrolled.)
12. Under treatment for graft versus host disease (GvHD). (GvHD cured subjects who had stopped immunosuppressive drugs for at least 1 month can be enrolled.)
13. Female subjects who are pregnant, breastfeeding or planning for pregnancy within 1 year after CAR-T cell infusion, or male subjects whose partners are planning for pregnancy within 1 year after CAR-T cell infusion;
14. Any conditions that would, in the investigator's assessment, increase risks in patients or interfere with the outcomes of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
BOR | 3 month
  Best Overall Response Rate

SECONDARY OUTCOMES:
ORR | 2 year
  Objective response rate
CR | 2 year
  Complete response rate
TTR | 3 month
  Time to response
DOR | 2 year
  Duration of response
EFS | 2 year
  Event-free survival
PFS | 2 year
  Progression-free survival
OS | 2 year
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided